CLINICAL TRIAL: NCT07375901
Title: The State of the Blood-Aqeous Barrier During Anti-Angiogenic Therapy in Patients With Exudative Age-Related Macular Degeneration
Brief Title: the Blood-Aqeous Barrier During Anti-Angiogenic Therapy in Exudative Age-Related Macular Degeneration
Acronym: BABAMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Filatov Institute of Eye Diseases and Tissue Therapy (Other)
Responsible Party: Principal Investigator, Andrii Korol, MD, PhD, Official Title: MD, PhD, DMedSc,Prof, The Filatov Institute of Eye Diseases and Tissue Therapy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0125U002070
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: AMD
Keywords: Age-related macular degeneration,laser flare photometry, anti-VEGF, aflibercept, brolucizumab,exudative
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group of aflibercept (Active Comparator): The first group (15 patients (17 eyes)) was administered intravitreal injections of 2 mg (0.05 mL) aflibercept.
  Interventions: Diagnostic Test: laser flare photometry before intravitreal injection
- Group of brolucizumab (Active Comparator): The second group (15 patients (16 eyes)) received 6 mg (0.05 mL) brolucizumab.
  Interventions: Diagnostic Test: laser flare photometry before intravitreal injection

INTERVENTIONS:
Diagnostic Test: laser flare photometry before intravitreal injection — The first group was administered intravitreal injections of 2 mg (0.05 mL) aflibercept The second group received 6 mg (0.05 mL) brolucizumab. Objectively measuring protein concentration in the aqueous humor using laser flare photometry (LFP).

SUMMARY:
To evaluate the status of the blood-aqueous barrier by objectively measuring protein concentration in the aqueous humor using laser flare photometry (LFP) in patients with exudative age-related macular degeneration (AMD) undergoing anti-angiogenic therapy.

DETAILED DESCRIPTION:
All patients were assigned to two groups. The first group was administered intravitreal injections of 2 mg (0.05 mL) aflibercept, while the second group received 6 mg (0.05 mL) brolucizumab. The regimen of treatment in both groups was treat-and-extend

ELIGIBILITY:
Inclusion Criteria: only primary, untreated patients with exudative AMD who were eligible for anti-VEGF therapy were included in the study. -

Exclusion Criteria:patients with hyperlipidemia, cardiac or renal insufficiency, ocular neoplasms, glaucoma, as well as those with corneal opacity within the optical zone or any inflammation of the studied eye that could lead to increased light-scattering intensity of protein molecules in the anterior chamber fluid, as measured by laser flare photometry, were excluded from the study.

-

Ages: 47 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
laser flare photometry values in the aqueous humor | 6-month
  Detection of protein concentration in the aqueous humor using laser flare photometry

SECONDARY OUTCOMES:
best-corrected visual acuity | 6-month
  the change in best-corrected visual acuity (BCVA)
central retinal thickness | 6-month
  central retinal thickness (CRT)

CONTACTS AND LOCATIONS:
Overall Officials: Andrii MD Korol, PhD, Principal Investigator — The Filatov Institute of Eye Diseases and Tissue Therapy
Locations (1):
- The Filatov Institute of Eye Diseases and Tissue Therapy, Odesa, Ukraine

IPD SHARING:
Plan to Share IPD: No